CLINICAL TRIAL: NCT02196064
Title: Hepatic Safety of Eviplera® in HIV/Hepatitis C (HCV)-Coinfected Patients Without HCV Treatment in the "The HEPAVIR HEPATIC SAFETY Cohort." hEPAtic Study.
Brief Title: Hepatic Safety of Eviplera® in HIV/Hepatitis C (HCV)-Coinfected Patients Without HCV Treatment in the "The HEPAVIR HEPATIC SAFETY Cohort."
Acronym: hEPAtic
Status: Completed | Type: Observational
Sponsor: Fundación Pública Andaluza Progreso y Salud (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Other Study IDs: hEPAtic
Record Dates: First submitted 2014-07-15; First posted 2014-07-21 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Human Immunodeficiency Virus (HIV) Hepatitis C Virus (HCV) Coinfected Subjects
Keywords: HIV HCV antiretroviral
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Safety of the three-drug combination TDF/FTC/RPV: A total of 176 patients will be included in this study, as well as 352 patients naive for RPV who initiated any ART that does not include RPV, who will serve as control group.

SUMMARY:
To evaluate the incidence of grade 3 or 4 transaminase elevations or grade 4 total bilirubin elevations (hepatic toxicity) during the first 48 weeks of antiretroviral therapy with the combination of rilpivirine (25mg), tenofovir (245mg) and emtricitabine (200mg), in a single-tablet regimen (Eviplera®) in human immunodeficiency virus (HIV)/hepatitis C virus (HCV)-coinfected subjects.

DETAILED DESCRIPTION:
This is a retrospective analysis of the prospective multicenter, observational "HEPAVIR HEPATIC SAFETY Cohort" (NCT01908660), in which the hepatic safety of the three-drug combination TDF/FTC/RPV will be assessed. A total of 176 patients will be included in this study, as well as 352 patients naive for RPV who initiated any ART that does not include RPV, who will serve as control group.

The main objective is to evaluate the incidence of grade 3 or 4 transaminase elevations or grade 4 total bilirubin elevations (hepatic toxicity) during the first 48 weeks of antiretroviral therapy with the combination of rilpivirine (25mg), tenofovir (245mg) and emtricitabine (200mg), in a single-tablet regimen (Eviplera®) in human immunodeficiency virus (HIV)/hepatitis C virus (HCV)-coinfected subjects.

Variables collected within in the cohort:

* Demographic variable: age, sex.
* Variables related to hepatitis C virus-infection: infection route, genotype, grade of hepatic fibrosis and method used for its determination, baseline Child-Pugh index in patients with cirrhosis, previous hepatic decompensations.
* Variables related to HIV-infection: CDC clinical category, HIV viral load, CD4 cell count, previous and new antiretroviral drugs.
* Blood test: AST, ALT platelets, cholesterol, bilirubin, gamma-glutamyltransferase, alkaline phosphatase, creatinine.
* Other variables: alcohol intake, self-reported adverse events, abnormal clinical findings.
* Cause of discontinuing antiviral when applicable.

Endpoints

1. Primary endpoint: Emergence of grade 3-4 TEs/grade 4 TBEs (hepatic toxicity) from baseline to week 48.
2. Secondary endpoints

   * Emergence of hepatic adverse events.
   * Drug interruptions due to liver toxicity.
   * Development of hepatic decompensations.
   * CD4 and viral load changes from baseline to week 48.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old.
* Chronic HIV-1 infection, as diagnosed on the basis of the presence of serum HIV antibodies detected by EIA and western-blot.
* Chronic HCV infection as proven by detecting HCV antibodies in plasma, as well as detectable plasma HCV-RNA by PCR.
* To start a new ART regimen during the study period.

Exclusion Criteria:

* Subjects with hepatotoxic events in the 2 months previous to Eviplera® treatment.
* Acute infections or uncontrolled chronic infection in the two months previous to Eviplera® treatment.
* Concomitant use of any drug with potential drug-drug interaction with Eviplera®.
* Documented resistance to study drugs.
* Concomitant therapy including anti-HCV agents, cytotoxic chemotherapy or immunosuppressors during Eviplera® treatment.
* Subjects taking part in any other clinical trial using an investigational product, with the exception of studies where the treatment studied have stopped for more than 12 weeks before Eviplera® treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 176 patients will be included in this study, as well as 352 patients naive for RPV who initiated any ART that does not include RPV, who will serve as control group.
Sampling Method: Probability Sample
Enrollment: 519 (Actual)
Dates: Start 2014-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Incidence of hepatic events | First 48 weeks of antiretroviral therapy
  Number of patients with grade 3 or 4 transaminase elevations or grade 4 total bilirubin elevations (hepatic toxicity) during the first 48 weeks of antiretroviral therapy with the combination of rilpivirine (25mg), tenofovir (245mg) and emtricitabine (200mg), in a single-tablet regimen (Eviplera®) in human immunodeficiency virus (HIV)/hepatitis C virus (HCV)-coinfected subjects.

SECONDARY OUTCOMES:
Comparison of hepatic events between exposed and unexposed to Eviplera® | First 48 weeks of antiretroviral therapy
  We evaluated the following parameters between subjets exposed and unexposed to Eviplera®
  * Incidence of hepatic toxicity
  * Incidence of hepatic adverse events.
  * Proportion of subjects who interrupt treatment due to liver toxicity according to Eviplera® exposure
  We will evaluated this parameters taking account the impact of baseline liver fibrosis/cirrhosis on liver toxicity.
Viral Kinetics and Immune response | 48 weeks of antiretroviral therapy
  Viral kinetics.- We compare the viral load between patients exposed and not exposed with Eviplera.
  Immune response.- We compare number of CD4 cells between patients exposed and not exposed with Eviplera

CONTACTS AND LOCATIONS:
Overall Officials: Juan Antonio Pineda Vergara, Study Chair — Hospital Universitario Virgen de Valme; Antonio Rivero Román, Study Chair — Hospital Universitario Reina Sofía; Dolores Merino Muñoz, Principal Investigator — Complejo Hospitalario de Especialidades Juan Ramón Jimenez; María José Rios Villega, Principal Investigator — Hospital Universitario Virgen Macarena; Francisco Téllez Pérez, Principal Investigator — Hospital La Línea de la Concepción; Inés Pérez Camacho, Principal Investigator — Hospital de Poniente; Antonio Collado Romacho, Principal Investigator — Complejo Hospitario Torrecárdenas; Josefa Ruiz Morales, Principal Investigator — Hospital Universitario Virgen de la Victoria; Marcial Delgado Fernández, Principal Investigator — Hospital Regional de Malaga; Leopoldo Muñoz Medina, Principal Investigator — Hospital Universitario San Cecilio; Francisco Vera Méndez, Principal Investigator — Hospital Santa María de Rosell; Nuria Espinosa Aguilera, Principal Investigator — Hospitales Universitarios Virgen del Rocío; Iganacio Santos Gil, Principal Investigator — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa; Juan González García, Principal Investigator — Hospital Universitario La Paz; Antonio Vergara de Campos, Principal Investigator — Hospital Universitario de Puerto Real; Juan Berenguer Berenguer, Principal Investigator — Hospital Universitario Gregorio Marañón; Federico Pulido Ortega, Principal Investigator — Hospital 12 de Octubre
Locations (1):
- Fundación Pública Andaluza Progreso y Salud, Seville, Sevilla, Spain